CLINICAL TRIAL: NCT05673252
Title: CERvical Cance The InFlammatory Index as a Predictor of risK Stratification:an Observational Study
Brief Title: CERvical Cancer The InFlammatory Index (CERTIFIKO)
Acronym: CERTIFIKO
Status: Recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Carlo Ronsini, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: 0035558/i
Record Dates: First submitted 2022-12-02; First posted 2023-01-06 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; neutrophil to lymphocyte ratio (NLR); lymphocyte to monocyte ratio (LMR); platelet to lymphocyte ratio (PLR)
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical cancer patients: The population is represented by women being admitted to the Gynecology Ward who are affected by cervical cancer.
  Interventions: Diagnostic Test: Venous blood sample; Procedure: biopsy

INTERVENTIONS:
Diagnostic Test: Venous blood sample — Blood chemistry tests: neutrophil;lymphocyte; monocyte; platelet counts
Procedure: biopsy — histopathology findings

SUMMARY:
Although significant advances in screening and treatment , cervical cancer is the fifth most common female cancer in Europe. Major prognostic factors for oncological outcome are used to categorise patients at high, intermediate and low risk groups and to define the type of radical hysterectomy according "Querleu-Morrow classification". The goal of this prospective observational study is to evaluate the association between several inflammatory markers and risk groups according European guidelines in women with cervical cancer Human Papillomavirus (HPV)-associated, in order to optimize the treatment.

DETAILED DESCRIPTION:
European guidelines have proposed a risk stratification of patients basing on oncological risk. The type of radical hysterectomy (extent of parametrial resection and type according Querleu-Morrow classification) should be based upon the presence of prognostic risk factors.Major prognostic factors for oncological outcome as tumour size, maximum stromal invasion, Lymphovascular space invasion (LVSI) are used to categorise patients at high, intermediate and low risk for treatment failure. The investigators want to identify additional parameters to better define risk profiles. Systemic inflammation indices such as neutrophil to lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR) and lymphocyte to monocyte ratio (LMR) have shown prognostic value in solid tumors and several inflammatory conditions. Therefore, the primary endpoint of the present study is to assess the role of systemic inflammatory indices and risk groups stratification in patients with early cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* At least 18-year-old patients.
* Patients histologically diagnosed with cervical cancer (squamous cell carcinoma or adenocarcinoma HPV- associated)
* Patients with (2018 FIGO) stage ≤ IB2 ("Early Cervical Cancer")
* Patients undergoing full-body CT-scan 30 days before enrollment.

Exclusion Criteria:

* Patients unfit to plead
* Patients with chronic inflammatory diseases (IBDs; rheumatic conditions)
* Synchronous tumors or cancer diagnosis in the previous 3 years
* Patients undergoing steroid therapy in the last 30 days prior to recruitment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histological diagnosis of cervical cancer undergoing surgical intervention who performed full-body CT-scan 30 days before enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2024-11-18 (Estimated); Study Completion 2024-11-18 (Estimated)

PRIMARY OUTCOMES:
Grading | 30 days after surgery
  Anatomic pathology report of cell anaplasia in the sampled tumor
Staging | 30 days after surgery
  Anatomic pathology report of extent to which the cancer has spread
Lymphovascular space invasion | 30 days after surgery
  Prognostic factor in cervical cancer
Histotype | 30 days after surgery
  Anatomic pathology report of tissue types of cancer
Tumor size | 30 days after surgery
  centimeters
Neutrophil-Lymphocyte Ratio (NLR) | 1 day previous surgery
  an absolute value obtained from the ratio of neutrophils to lymphocytes
Platelet-lymphocyte ratio(PLR) | 1 day previous surgery
  an absolute value obtained from the ratio of platelets to lymphocytes
Lymphocyte-monocyte Ratio (LMR) | 1 day previous surgery
  an absolute value obtained from the ratio of lymphocytes to monocytes

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Ronsini, MD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Università degli Studi della Campania Luigi Vanvitelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes